CLINICAL TRIAL: NCT02291640
Title: Coparison of Miller and CoPilot Laryngoscopes for Intubation by Nurses During Child Chest Compression. A Manikin Study
Brief Title: Pediatric Intubation Among Nursing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/16
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest; Intubation, Endotracheal
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child ETI with chest compressions (Experimental): endotracheal intubation (ETI) during child mannikin resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: MIL; Device: CoPilot
- Child ETI without chest compressions (Experimental): Endotracheal intubation of child mannikin during resuscitation without chest compressions.
  Interventions: Device: MIL; Device: CoPilot

INTERVENTIONS:
Device: MIL — direct laryngoscopy
  Other Names: Miller laryngoscope
Device: CoPilot — video laryngoscopy
  Other Names: CoPilot VideoLaryngoscope

SUMMARY:
The aim of this study was to compare time, success rates of video laryngoscope and direct laryngoscope for the emergency intubation with an immobilized cervical spine in a standardized pediatric manikin model.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in nursing

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices.

SECONDARY OUTCOMES:
Time to intubation | 1 day
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.If the examinee failed at all attempts, the case was excluded from the time calculations.

OTHER OUTCOMES:
Cormack-Lehan scale | 1 day
  self reported Cormack-Lehan scale during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland